CLINICAL TRIAL: NCT04672499
Title: A Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of Miricorilant Tablet Formulations Following Single and Multiple Oral Doses in Healthy Participants
Brief Title: Single and Multiple Dose Study of Miricorilant (CORT118335) Tablet Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CORT118335-853; 2019-004655-36 (EudraCT Number)
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Healthy
MeSH Terms: interventions — CORT118335

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Cohort 1: Miricorilant 900 mg (Regimen A1) (Experimental): Participants will receive a single oral dose of miricorilant 900 mg (3 X 300 mg) after breakfast on Day 1. Cohort 1 treatment will be randomized and open label.
  Interventions: Drug: Miricorilant 300 mg tablets
- Cohort 1: Miricorilant 300 mg (Regimen A2) (Experimental): Participants will receive a single oral dose of miricorilant 300 mg (2 X 150 mg) after breakfast on Day 1. Cohort 1 treatment will be randomized and open label.
  Interventions: Drug: Miricorilant 150 mg tablets
- Cohort 2: Miricorilant (Regimen B1 and B2) (Experimental): Participants will receive a single oral dose of miricorilant 900 mg (6 X 150 mg) after breakfast on Day 1 (Regimen B1). After a minimum 7-day washout, participants will receive miricorilant 900 mg (6 X 150 mg) qd for 14 days (Regimen B2). Day 1 treatment in Regimen B2 will be in the fasted state; the remaining doses will follow breakfast. Cohort 2 treatments will be randomized and blinded.
  Interventions: Drug: Miricorilant 150 mg tablets
- Cohort 2: Placebo (Regimen B1 and B2) (Placebo Comparator): Participants will receive a single oral dose of placebo matching miricorilant 900 mg (6 X 150 mg) after breakfast on Day 1 (Regimen B1). After a minimum 7-day washout, participants will receive placebo matching miricorilant 900 mg (6 X 150 mg) qd for 14 days (Regimen B2). Day 1 treatment in Regimen B2 will be in the fasted state; the remaining doses will follow breakfast. Cohort 2 treatments will be randomized and blinded.
  Interventions: Drug: Placebo 150 mg tablets
- Cohort 3: Miricorilant (Regimen C1 and C2) (Experimental): Participants will receive two oral doses (morning and evening) of miricorilant 1350 mg (9 X 150 mg) after a meal on Day 1 (Regimen C1). After a minimum 7-day washout, participants will receive miricorilant 750 mg (5 X 150 mg) after breakfast for 14 days and miricorilant 600 mg (4 X 150 mg) in the evening after a meal for 13 days (Regimen C2). Cohort 3 treatments will be randomized and blinded.
  Interventions: Drug: Miricorilant 150 mg tablets
- Cohort 3: Placebo (Regimen C1 and C2) (Placebo Comparator): Participants will receive two oral doses (morning and evening) of placebo matching miricorilant 1350 mg (9 X 150 mg) after a meal on Day 1 (Regimen C1). After a minimum 7-day washout, participants will receive placebo matching miricorilant 750 mg (5 X 150 mg) after breakfast for 14 days and placebo matching miricorilant 600 mg (4 X 150 mg) in the evening after a meal for 13 days (Regimen C2). Cohort 3 treatments will be randomized and blinded.
  Interventions: Drug: Placebo 150 mg tablets

INTERVENTIONS:
Drug: Miricorilant 300 mg tablets — Miricorilant 300 mg tablets for oral administration
  Other Names: CORT118335
  Arms: Cohort 1: Miricorilant 900 mg (Regimen A1)
Drug: Miricorilant 150 mg tablets — Miricorilant 150 mg tablets for oral administration
  Other Names: CORT118335
  Arms: Cohort 1: Miricorilant 300 mg (Regimen A2); Cohort 2: Miricorilant (Regimen B1 and B2); Cohort 3: Miricorilant (Regimen C1 and C2)
Drug: Placebo 150 mg tablets — Placebo to match miricorilant 150 mg tablets for oral administration
  Arms: Cohort 2: Placebo (Regimen B1 and B2); Cohort 3: Placebo (Regimen C1 and C2)

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetics (PK) of miricorilant (CORT118335) tablet formulations following single and multiple oral administration in healthy participants.

DETAILED DESCRIPTION:
Cohort 1 will evaluate safety, tolerability, and PK of single doses of a 150-mg and a new 300-mg tablet formulation of miricorilant. Cohort 1 treatment will be randomized and open label.

Optional Cohorts 2 and 3 will evaluate single- and repeated-dose administration of miricorilant using a formulation, dose, and dose-regimen determined after interim evaluation of PK and safety data from previous cohorts. Cohort 2 and 3 treatments will be randomized, blinded, and placebo controlled.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 30.0 kg/m^2
* Must agree to adhere to the contraception requirements
* Additional criteria apply.

Exclusion Criteria:

* Received any investigational medicinal product in a clinical research study within the last 90 days
* Male participants who have pregnant or lactating partners
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption: a confirmed positive alcohol breath test at screening or admission
* Current smokers and those who have smoked or used e-cigarettes or nicotine replacement products within the last 6 months
* Females of childbearing potential including those who are pregnant or lactating (all female subjects must have a negative serum pregnancy test at screening and a negative urine pregnancy test at admission)
* Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the Investigator
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Active renal and/or hepatic disease
* History of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, chronic respiratory, neurological or psychiatric disorder, as judged by the Investigator
* Any form of cancer within the last 2 years (exceptions apply)
* History and/or symptoms of adrenal insufficiency
* Regularly consumes liquorice or other glycyrrhetic acid derivatives
* History of clinically significant gastrointestinal disease
* Currently using glucocorticoids or have a history of systemic glucocorticoid use within the last 12 months or 3 months for inhaled products
* Presence or history of clinically significant allergy requiring treatment
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Taking, or have taken, any prescribed, over-the-counter drug (other than up to 4 g per day paracetamol) or vitamins/herbal remedies within 14 days. Exceptions may apply on a case by case basis
* Additional criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with One or More Adverse Events | Up to 7±2 days after the last dose (up to approximately Day 9 for Cohort 1 and up to approximately Day 23 for Cohorts 2 and 3)
Percentage of Participants with One or More Serious Adverse Events | Up to 7±2 days after the last dose (up to approximately Day 9 for Cohort 1 and up to approximately Day 23 for Cohorts 2 and 3)
Percentage of Participants Discontinued from the Study due to an Adverse Event | Up to 7±2 days after the last dose (up to approximately Day 9 for Cohort 1 and up to approximately Day 23 for Cohorts 2 and 3)

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK) of Miricorilant: Elapsed Time from Dosing at which the Analyte was First Quantifiable in a Concentration vs Time Profile (tlag) | Single-dose regimens: before dosing and at pre-specified time points up to 72 hours after dosing (Day 4)
Plasma PK of Miricorilant: Maximum Observed Concentration (Cmax) | Single-dose regimens: before dosing and at pre-specified time points up to 72 hours after dosing (Day 4); Repeated-dose regimens: before dosing and at pre-specified time points up to 72 hours after final dose (Day 17)
Plasma PK of Miricorilant: Time from Dosing at which Cmax was Apparent (Tmax) | Single-dose regimens: before dosing and at pre-specified time points up to 72 hours after dosing (Day 4); Repeated-dose regimens: before dosing and at pre-specified time points up to 72 hours after final dose (Day 17)
Plasma PK of Miricorilant: Apparent Elimination Half-life (t1/2) | Single-dose regimens: before dosing and at pre-specified time points up to 72 hours after dosing (Day 4); Repeated-dose regimens: before dosing and at pre-specified time points up to 72 hours after final dose (Day 17)
Plasma PK of Miricorilant: Area Under the Curve from Time Zero to the Last Measurable Concentration (AUC0-last) | Single-dose regimens: before dosing and at pre-specified time points up to 72 hours after dosing (Day 4)
Plasma PK of Miricorilant: Area Under the Curve from Time Zero to 24 Hours Postdose (AUC0-24) | Repeated-dose regimens: before dosing and at pre-specified time points up to 72 hours after final dose (Day 17)

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No